CLINICAL TRIAL: NCT01361568
Title: A Multi-Center, Double-Randomized, Double Blind, Placebo Controlled Study to Evaluate the Analgesic Efficacy and Safety of Intravenous CR845 Dosed Preoperatively and Postoperatively in Patients Undergoing a Laparoscopic Hysterectomy
Brief Title: Study to Evaluate Analgesic Effect of IV Administration of Kappa Agonist CR845 For Hysterectomy Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR845 CLIN2002
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Postoperative Pain
Keywords: pain; acute pain; visceral pain; kappa agonist; opioid analgesics; peripheral nervous system agents; physiological effects of drugs; surgery; hysterectomy; post-operative; post-operative complications
MeSH Terms: conditions — Pain, Postoperative; Pain; Acute Pain; Visceral Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CR845 (Experimental): Peripheral kappa opioid receptor agonist
  Interventions: Drug: CR845
- Placebo (Placebo Comparator): Matched Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CR845 — Single i.v. dose (0.04 mg/kg) administered preoperatively
  Other Names: Preoperative Active Dose
  Arms: CR845
Drug: Placebo — Single i.v. dose administered preoperatively
  Other Names: Preoperative Placebo Dose
  Arms: Placebo
Drug: CR845 — Single i.v. dose (0.04 mg/kg) administered postoperatively for pain
  Other Names: Postoperative Active for Pain
  Arms: CR845
Drug: Placebo — Single i.v. dose administered postoperatively for pain
  Other Names: Postoperative Placebo for Pain
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to determine if CR845 is effective in treating the pain associated with a laparoscopic hysterectomy.

DETAILED DESCRIPTION:
Currently, the most widely used drugs to treat pain after surgery are opiates, such as morphine. Morphine works mainly by activating one of several types of opiate receptors that control some of our pain sensation - the so-called mu opiate receptors. These receptors are located in many areas of the brain and also outside of the brain. By activating these receptors, morphine provides significant pain relief, but also causes side effects that limit its use. Some of these side effects include: respiratory depression or arrest (slowed or stopped breathing), sedation (a state of calmness or extreme relaxation), euphoria (an exaggerated feeling of physical and mental well-being), constipation, nausea, vomiting, and drug addiction.

In order to avoid the side effects of morphine and other mu opiates, the present experimental drug CR845 was designed to work at a different type of opiate receptor - called kappa - that can also provide pain relief, by acting on sensory nerves outside the brain. CR845 was designed to penetrate the brain much less than other opiate drugs, which should result in pain relief similar to that of morphine, but with fewer side effects. Because CR845 activates kappa receptors instead of mu receptors, the side effects are different than with a morphine-type drug. In particular, kappa opiates, such as CR845, do not cause respiratory depression or arrest, euphoria, constipation, drug tolerance, physical drug dependence or drug addiction. For these reasons, CR845 may present a distinct advantage over other opiates that are currently used for pain relief and post-operative pain in particular.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent prior to any study procedures;
* Able to communicate clearly with the Investigator and staff;
* Female between 21 and 65 years of age, inclusive;
* Scheduled for elective laparoscopic hysterectomy under general anesthesia;
* Negative result on serum pregnancy test at screening and negative urine pregnancy test at Baseline (for women of child-bearing potential only) and not currently breast feeding, or planning to do so within 30 days of dosing;
* Negative urine drug screen for drugs of abuse at Screening and at Baseline;
* American Society of Anesthesiologists (ASA) risk class of I to III;
* Body mass index (BMI) between 17 and 40 inclusive.

Exclusion Criteria:

* Has known allergies to opioids, or hypersensitivity to other materials (such as infusion line) or medications to be used in the study;
* Has a known or suspected history of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)-diagnosed alcohol, opiate or other drug abuse or dependence within 12 months prior to screening;
* Is unable to refrain from alcohol consumption for a period beginning 24 hours prior to surgery through the end of the Treatment Period;
* Is scheduled to undergo a hysterectomy that will utilize any type of robotic technology and/or a concomitant surgical procedure that would produce a significantly greater degree of surgical trauma than the laparoscopic hysterectomy or laparoscopic assisted vaginal hysterectomy alone;
* Has taken non-opioid analgesics (including cyclooxygenase-2 [COX-2] inhibitors) or nonsteroidal anti-inflammatory drugs (NSAIDs) within 12 hours of the Baseline assessments;
* Has taken any opioid analgesics or used systemic steroids within 4 days of surgery OR has previously used opiates chronically for a period of ≥3 months;
* Has used antipsychotics, antiepileptics, sedatives, hypnotics, or antianxiety agents, selective serotonin reuptake inhibitors (SSRIs), tricyclic antidepressants for < 30 days prior to surgery or had a dose change within the previous 30 days;
* Has taken any prescription or over-the-counter medication within 3 days prior to surgery that, in the opinion of the Investigator, is expected to confound the analgesic response;
* Has taken herbal agents or nutraceuticals (i.e., chaparral, comfrey, germander, gin bu huan, kava, pennyroyal, skullcap, St. John's wort, or valerian) 7 days prior to surgery;
* In the opinion of Investigator shows clinical signs of hypovolemia;
* Has an oxygen saturation < 92% on room air at Screening or prior to receiving the first infusion of study drug;
* Has any history of clinically significant cardiovascular disease,
* Has a clinically significant abnormal electrocardiogram (ECG) or a history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome);
* Has a history of any serious medical conditions that in the opinion of the Investigator would preclude study participation;
* Has serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, or gamma glutamyl transferase (GGT) >2.5 x the upper limit of normal (ULN) at screening;
* Has bilirubin, blood urea nitrogen (BUN), or creatinine >1.5 x the reference ULN at Screening;
* Has abnormally low hemoglobin < 10 mg/dl at Screening;
* Has serum sodium levels > 146 mmol/L at Screening;
* Has impaired renal function (creatinine clearance [CrCl] < 50 ml/min) at Screening;
* Has a positive test for human immunodeficiency virus (HIV) or known history of HIV infection;
* Has received another investigational drug within 30 days of scheduled surgery;
* Has a significant chronic pain condition in areas unrelated to the operative site at the time of Screening that in the Investigator's opinion could confound the interpretation of study results

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tong-Joo Gan, MD, MHS, Principal Investigator — Duke University
Locations (18):
- United States (18):
  - Shoals Clinical Research Associates, Florence, Alabama
  - Horizon Research Group, Mobile, Alabama
  - Wilmax, Mobile, Alabama
  - Drug Research and Analysis Corp, Montgomery, Alabama
  - Shoals Medical Trials, INC, Sheffield, Alabama
  - Precision Clinical Trials, Phoenix, Arizona
  - Woodland Healthcare California Clinical Research, Inc, Davis, California
  - Olive View-UCLA Medical Center, Sylmar, California
  - Visions Clinical Research, Boynton Beach, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - University of Miami, Dept of, Miami, Florida
  - Cypress Medical Research, Wichita, Kansas
  - Cooper University Hospital, Camden, New Jersey
  - Duke University, Durham, North Carolina
  - Ohio State University Medical, Dept of Anesthesia, Columbus, Ohio
  - Palmetto Clinical Research,, Greenville, South Carolina
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - Texas Health Care, PLLC, Fort Worth, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo-Placebo: Placebo administered both preoperatively and postoperatively
- Placebo-CR845: Placebo administered preoperatively and CR845 administered postoperatively
- CR845-CR845: CR845 administered both preoperatively and postoperatively
- CR845-Placebo: CR845 administered preoperatively and placebo administered postoperatively
- CR845-No Postoperative Treatment: CR845 administered preoperatively and no study drug administered postoperatively
- Placebo-No Postoperative Treatment: Placebo administered preoperatively and no study drug administered postoperatively
Period: Overall Study
Arm/Group | Placebo-Placebo | Placebo-CR845 | CR845-CR845 | CR845-Placebo | CR845-No Postoperative Treatment | Placebo-No Postoperative Treatment
Started | 71 | 71 | 20 | 21 | 7 | 13
Completed | 69 | 70 | 20 | 21 | 6 | 11
Not Completed | 2 | 1 | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-Placebo | Placebo-CR845 | CR845-CR845 | CR845-Placebo | CR845-No Postoperative Treatment | Placebo-No Postoperative Treatment | Total
Number analyzed (Participants) | 71 | 71 | 20 | 21 | 7 | 13 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 71 | 70 | 20 | 21 | 7 | 13 | 202
  >=65 years | 0 | 1 | 0 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (8.60) | 44.3 (9.69) | 43.8 (7.14) | 40.0 (6.88) | 55.9 (7.84) | 45.3 (7.93) | 43.7 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 71 | 20 | 21 | 7 | 13 | 203
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 71 | 71 | 20 | 21 | 7 | 13 | 203

OUTCOME MEASURES:

1. Primary Outcome: Total Morphine Consumption in the First 24 Hours Following Postoperative Study Drug Treatment
Time Frame: 24 hours
Population: The primary analysis included all patients in the modified Intent-to-Treat (mITT) population who re-randomized in the postoperative period, where time 0 was the start time of the postoperative study drug infusion.
Measure: Mean (Standard Error); unit: mg
Arm/Group | Placebo-Placebo | Placebo-CR845 | CR845-CR845 | CR845-Placebo
Number analyzed (Participants) | 71 | 71 | 20 | 21
mg | 21.9 (1.89) | 17.6 (1.65) | 13.9 (2.20) | 19.8 (3.03)
Statistical Analysis 1: Comparison: Placebo-Placebo vs CR845-CR845; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -7.96, 95% CI 2-sided [-15.14 to -0.78], Standard Error of Mean 3.64

2. Secondary Outcome: Summed Pain Intensity Difference From 0-24 Hours (SPID 0-24) Following Postoperative Study Drug Treatment Using Last Observation Carried Forward (LOCF)
Description: Patients reported their pain intensity using a visual analogue scale (VAS) from 0 to 100 mm, where 0 mm represented "No Pain" and 100 mm represented the "Worst Pain You Can Imagine". SPID 0-24 represents the cumulative time-weighted sum of the pain intensity difference (PID) scores between each assessment timepoint following the postoperative administration of study drug (i.e. 0 to 15 min, 15 to 30 min, etc.) over 24 hours. Pain intensity assessments were measured at baseline (entry pain score), then at 15, 30, 45, 60, 90, 120, 150, 180, 240, 360, 480, 720, 960, and 1440 minutes after the start of the infusion of study drug following surgery.
  Negative SPID values represent a decrease in pain intensity (i.e. lower values indicate a greater reduction in pain).
Time Frame: 0 to 24 hours
Population: The analysis included all patients in the modified Intent-to-Treat (mITT) population who re-randomized in the postoperative period, where time 0 was the start time of the postoperative study drug infusion, and did not have a missing baseline pain intensity score.
Measure: Mean (Standard Error); unit: units on a scale * hours
Arm/Group | Placebo-Placebo | Placebo-CR845 | CR845-CR845 | CR845-Placebo
Number analyzed (Participants) | 71 | 71 | 20 | 19
units on a scale * hours | -413.1 (67.8) | -643.2 (58.11) | -833.1 (124.8) | -673.5 (152.36)
Statistical Analysis 1: Comparison: Placebo-Placebo vs CR845-CR845; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = -420, Standard Error of Mean 139.16
Statistical Analysis 2: Comparison: Placebo-Placebo vs Placebo-CR845; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -230.1, Standard Error of Mean 92.26
Statistical Analysis 3: Comparison: Placebo-Placebo vs CR845-Placebo; Test type: Superiority or Other; p = 0.068, t-test, 2 sided; Mean Difference (Final Values) = -260.4, Standard Error of Mean 141.99

3. Secondary Outcome: Morphine Consumption Following Postoperative Study Drug Treatment in the 2-24 Hour Period After Recovery in the Post-Anesthesia Care Unit (Post-PACU)
Time Frame: 2 to 24 hours (post-PACU)
Population: The analysis included all patients in the modified Intent-to-Treat (mITT) population who re-randomized in the postoperative period, where time 0 was the start time of the postoperative study drug infusion. Morphine consumption was calculated for the 2-24 hour period, after patients were transferred out of the PACU.
Measure: Mean (Standard Error); unit: mg
Arm/Group | Placebo-Placebo | Placebo-CR845 | CR845-CR845 | CR845-Placebo
Number analyzed (Participants) | 71 | 71 | 20 | 21
mg | 14.38 (1.35) | 11.07 (1.17) | 7.99 (2.03) | 11.33 (2.11)
Statistical Analysis 1: Comparison: Placebo-Placebo vs CR845-CR845; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Least Squares Mean Difference = -6.39, Standard Error of Mean 2.63
Statistical Analysis 2: Comparison: Placebo-Placebo vs Placebo-CR845; Test type: Superiority or Other; p = 0.059, Mixed Models Analysis; Least Squares Mean Difference = -3.31, Standard Error of Mean 1.74

4. Secondary Outcome: Total Pain Relief Within the First 2 Hours (TOTPAR 0-2) Following Postoperative Study Drug Treatment Using LOCF
Description: Patients reported their pain relief using a 5-point categorical scale of 0 to 4 (0 = No Relief, 1 = A Little Relief, 2 = Some Relief, 3 = A Lot of Relief and 4 = Complete Relief). TOTPAR 0-2 was represents the cumulative time-weighted sum of the pain relief (PR) scores between each assessment timepoint following the postoperative administration of study drug (i.e. 15 to 30 min, 30 to 45 min, etc.) over the first 2 hours. Pain relief assessments were measured at 15, 30, 45, 60, 90, 120 minutes after the start of the infusion of study drug following surgery.
  Positive TOTPAR values represent an increase in pain relief.
Time Frame: 0 to 2 hours
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale * hours
Arm/Group | Placebo-Placebo | Placebo-CR845 | CR845-CR845 | CR845-Placebo
Number analyzed (Participants) | 71 | 71 | 20 | 19
units on a scale * hours | 1.4 (0.16) | 2.1 (0.19) | 2.4 (0.48) | 1.5 (0.40)
Statistical Analysis 1: Comparison: Placebo-Placebo vs CR845-CR845; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [0.22 to 1.82], Standard Error of Mean 0.41
Statistical Analysis 2: Comparison: Placebo-Placebo vs Placebo-CR845; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [0.11 to 1.17], Standard Error of Mean 0.27

5. Secondary Outcome: Global Evaluation Responder Analysis
Description: Responders = Excellent or Very Good; Non-Responders = Fair or Poor. Patient who reported a score of "Good" were not included in the analysis as the midpoint cannot be unambiguously assigned for a binary outcome measurement.
Time Frame: At 24 hours
Population: The responder analysis included all patients in the modified Intent-to-Treat (mITT) population and compared patients that received any dose of CR845 (preoperatively and/or postoperatively) to patients that only received placebo.
Measure: Number; unit: Responder Count
Groups:
- Placebo: Patients administered placebo only either preoperatively and/or postoperatively
- CR845: Patients administered CR845 either preoperatively and/or postoperatively
Arm/Group | Placebo | CR845
Number analyzed (Participants) | 55 | 90
Responder Count | 27 | 68
Statistical Analysis 1: Comparison: Placebo vs CR845; Test type: Superiority or Other; p = 0.001, Chi-squared; Degrees of freedom (df = 1)

6. Secondary Outcome: Total Number of Patients Reporting At Least One Episode of Nausea
Time Frame: Up to 24 hours
Population: All patients in the modified Intent-to-Treat (mITT) population and compared patients that received any dose of CR845 (preoperatively and/or postoperatively) to patients that only received placebo.
Measure: Number; unit: percentage of patients
Groups:
- Placebo: Patients administered placebo only, either preoperatively and/or postoperatively
Arm/Group | Placebo | CR845
Number analyzed (Participants) | 84 | 119
percentage of patients | 51.2 | 26.1
Statistical Analysis 1: Comparison: Placebo vs CR845; Test type: Superiority or Other; p < 0.001, Fisher Exact

7. Secondary Outcome: Total Number of Patients Reporting At Least One Episode of Vomiting
Time Frame: Up to 24 hours
Population: as for outcome 6
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | CR845
Number analyzed (Participants) | 84 | 119
percentage of patients | 8.3 | 1.7
Statistical Analysis 1: Comparison: Placebo vs CR845; Test type: Superiority or Other; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the time the patient received her first dose of study drug through the Follow-up Visit.
Arm/Group | Placebo-Placebo | Placebo-CR845 | CR845-CR845 | CR845-Placebo | CR845-No Postoperative Treatment | Placebo-No Postoperative Treatment
Serious Adverse Events (participants affected / at risk) | 0/71 | 6/71 | 3/20 | 0/21 | 3/7 | 1/13
Other Adverse Events (participants affected / at risk) | 59/71 | 62/71 | 19/20 | 15/21 | 7/7 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-Placebo (N=71) | Placebo-CR845 (N=71) | CR845-CR845 (N=20) | CR845-Placebo (N=21) | CR845-No Postoperative Treatment (N=7) | Placebo-No Postoperative Treatment (N=13)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Sodium Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic Adhesions (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-Placebo (N=71) | Placebo-CR845 (N=71) | CR845-CR845 (N=20) | CR845-Placebo (N=21) | CR845-No Postoperative Treatment (N=7) | Placebo-No Postoperative Treatment (N=13)
Nausea (Gastrointestinal disorders) | 38 (39) | 26 (26) | 9 (9) | 5 (5) | 1 (1) | 5 (5)
Flatulence (Gastrointestinal disorders) | 18 (18) | 9 (9) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 11 (11) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal Dilatation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 14 (14) | 18 (18) | 4 (4) | 5 (5) | 2 (2) | 5 (5)
Hypertension (Vascular disorders) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 10 (10) | 9 (9) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 4 (4) | 0 (0)
Hypoaesthesia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysstasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Sodium Increased (Investigations) | 0 (0) | 12 (12) | 7 (7) | 8 (8) | 1 (1) | 0 (0)
Blood Chloride Increased (Investigations) | 0 (0) | 8 (8) | 6 (6) | 8 (8) | 1 (1) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Airway Peak Pressure Increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine Output Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Retension (Renal and urinary disorders) | 6 (7) | 8 (9) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Bladder Spasm (Renal and urinary disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 7 (7) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Incisional Site Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental Status Change (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensation of Pressure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscule Spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diploplia (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast Tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days